CLINICAL TRIAL: NCT05187208
Title: A Phase IV Open-label, Multicenter Study of Niraparib as Maintenance Therapy in BRCA Wild-type, Newly Diagnosed Advanced Ovarian Cancer Patients in Korea
Brief Title: PARP Inhibitor Oral Maintenance in Low-Risk Ovarian Cancer
Acronym: POLO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Yonsei University (Other); Asan Medical Center (Other); Samsung Medical Center (Other); Takeda (Industry)
Responsible Party: Principal Investigator, Jae-Weon Kim, Seoul National University Hospital, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCR-2021-200106
Record Dates: First submitted 2021-12-19; First posted 2022-01-11 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Epithelial Ovarian Cancer; Ovarian Cancer; Ovarian Cancer Stage III; Ovarian Cancer Stage IV
Keywords: Epithelial Ovarian Cancer; Ovarian Cancer; Maintenance; Molecular Targeted Therapy
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Ovarian Neoplasms | interventions — niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): BRCA1/2 wild-type, advanced-stage, low-risk, primary ovarian cancer patients (high-grade serous or high-grade endoemtrioid)
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib — Niraparib 200mg or 300mg (once daily [QD])*
  *The recommended starting dosage of niraparib is 200mg QD. For patients who weigh ≥77 kg and have baseline platelet count ≥150,000/μL, the recommended starting dosage is 300 mg QD.

SUMMARY:
This study is the phase IV, open-label, clinical trial to determine the efficacy of niraparib maintenance therapy in BRCA1/2 wild-type, advanced-stage, low-risk, primary ovarian cancer patients.

DETAILED DESCRIPTION:
This study is a phase IV, open-label, clinical trial to determine the efficacy of niraparib maintenance therapy in BRCA1/2 wild-type, advanced-stage, low-risk, primary ovarian cancer patients. The study will assess the effectiveness of progression-free survival (12 months PFS rate) as determined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. The subject will be treated up to three years or until disease progression as below:

Niraparib 200mg or 300mg (once daily [QD])*

*The recommended starting dosage of niraparib is 200mg QD. For patients who weigh ≥77 kg and have baseline platelet count ≥150,000/μL, the recommended starting dosage is 300 mg QD.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has histologically confirmed diagnosis of FGIO stage III-IV high-grade serous or high-grade endometrioid ovarian cancer, primary peritoneal cancer, or fallopian tube cancer will be enrolled in this study.
2. Participant has confirmed as both germline and somatic BRCA1/2 wild-type by institution's test.
3. Participant has no visible residual tumor after primary cytoreductive surgery (or optimally debulked) and has responded to the postoperative platinum-based combination chemotherapy (complete or partial response), remains in response, and is enrolled on study within 12 weeks of completion of the last platinum regimen
4. Participant who is able to provide tumor slides obtained during cytoreductive surgery for a prospective examination of the homologous recombination deficiency (HRD).
5. Female participants who are at least 20 years of age on the day of signing informed consent with
6. Participant has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1, as assessed within 10 days prior to enrollment.
7. Participant is eligible to participate if she is not pregnant (see Appendix 2), not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 2 OR
   2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 2 during the treatment period and for at least 180 days following the last dose of niraparib.
8. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial. The participant may also provide consent for future biomedical research; however, the participant may participate in the main study without participating in future biomedical research.
9. Participant has adequate organ function as defined in the following table (Table 1).; all screening laboratory tests should be performed within 10 days prior to the start of study treatment.

Exclusion Criteria:

1. Participant has mucinous, germ cell, or borderline tumor of the ovary.
2. Participant receives neoadjuvant chemotherapy before cytoreductive surgery.
3. Participant has a visible residual tumor after primary cytoreductive surgery.
4. Participant receives bevacizumab with front-line platinum-based combination chemotherapy.
5. Participant has a history of non-infectious pneumonitis that required treatment with steroids or currently has pneumonitis.
6. Participant either has myelodysplastic syndrome (MDS)/ acute myeloid leukemia (AML) or has features suggestive of MDS/AML.
7. Participant has a known additional malignancy that is progressing or has required active treatment within the past 2 years.

   Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ, endometrial carcinoma) that have undergone potentially curative therapy are not excluded.

   Note: Participants with synchronous primary endometrial cancer or a past history of primary endometrial cancer that met the following conditions are not excluded: Stage not greater than IA: no more than superficial myometrial invasion.
8. Drainage of ascites during the last 2 cycles of last chemotherapy.
9. Palliative radiotherapy within 1 week encompassing >20% of the bone marrow.
10. Persistent >grade 2 toxicity from prior cancer therapy.
11. Symptomatic uncontrolled brain or leptomeningeal metastases. A scan to confirm the absence of brain metastases is not required. Patients with spinal cord compression may be considered if they have received definitive treatment for this and evidence of clinically stable disease for 28 days.
12. Major surgery within 3 weeks of starting the study or patient has not recovered from any effects of any major surgery.
13. Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease, or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent.
14. History or current evidence of any condition, therapy, or lab abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study treatment or is not in the best interest of the patient to participate.
15. Patient is pregnant or breast feeding, or expecting to conceive children within the projected duration of the study treatment.
16. Immunocompromised patients.
17. Patients with known active hepatic disease (i.e., Hepatitis B or C).

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (12 month PFS rate) | 12 months
  To determine the clinical effectiveness of the study treatment assessed using progression free survival (12 months) according to RECIST v1.1 criteria (Investigator determined)

SECONDARY OUTCOMES:
Progression-free survival | 36 months
Overall survival (OS) | 36 months
Time to second objective disease progression (PFS2) | 36 months
Time to second subsequent treatment (TSST) | 36 months

OTHER OUTCOMES:
12 month PFS rate by homologous recombination deficiency (HRD) status | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Weon Jae-Weon, MD, PhD, Principal Investigator — Seoul National University Hpospital

IPD SHARING:
Plan to Share IPD: Undecided